CLINICAL TRIAL: NCT03953352
Title: Evaluation of the Automatic Deformable Recontouring on the Daily MVCT for Head and Neck Cancer Adaptive Radiotherapy
Acronym: GIRAFE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study cancelled
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19VADS01
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Cancer
Keywords: Adaptive radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy treatment (Other)
  Interventions: Other: Helical intensity-modulated radiotherapy (IMRT)

INTERVENTIONS:
Other: Helical intensity-modulated radiotherapy (IMRT) — Helical intensity-modulated radiotherapy (35 fractions, 5 fractions per week) will be administered during 7 weeks: 2 Gy per fraction on tumor and 1.6 Gy per fraction on bilateral lymph node areas.

SUMMARY:
This trial is a prospective, monocentric study aiming to evaluate an adaptive radiotherapy method (automatic deformable recontouring on the daily MVCT (MegaVoltage Computerized Tomography)) using the Precise ART™ software in patients with head and neck cancer.

Patients will receive helical intensity-modulated radiotherapy (IMRT) according to the standard recommendations (35 fractions during 7 weeks). Radiotherapy will include daily repositioning MVCT.

For the study, patients will undergo 4 intermediate re-planning CT-scan (without injection of intravenous contrast agent) at week 3, week 4, week 5 and week 6 of treatment.

3 recontouring modalities will be evaluated for the study:

* Manuel recontouring (standard method)
* Precise ART™ deformed contours
* Precise RTX™ deformed contours

The total duration of the study for each patient will be 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patient with histologically proven locally advanced head and neck cancer (Oropharynx, hypopharynx, larynx, nasopharynx, oral cavity, sinuses, nasal cavities, ethmoid sinus, cavum, salivary glands)
3. Cancer with nodal involvement (at least T3 or involved node >2 cm)
4. Eastern Cooperative Oncology Group performance status 0 or 1
5. No previous curative treatment for head and neck cancer (surgery and/or radiotherapy and/or chemotherapy)
6. Indication of exclusive radiotherapy (+/- chemotherapy) validated in multidisciplinary meeting
7. Patient affiliated to the french social security system.
8. Patient must provide written informed consent prior to inclusion in the study and any study-specific procedure.

Exclusion Criteria:

1. Patient with metastatic cancer
2. Eastern Cooperative Oncology Group performance status ≥ 2 (due to comorbidities)
3. Patient with recurrent disease
4. Patient who required urgent surgical treatment
5. Contraindications to radiotherapy
6. History of cancer within 5 years
7. Patient already included in another therapeutic trial
8. Pregnant or breastfeeding women
9. Any psychological, familial, geographical or sociological condition potentially preventing the medical follow-up and/or study procedures
10. Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with Dice Similarity Coefficient (DSC) of the volumes of left and right parotid gland superior to 0.85 (DSC > 0.85) | 7 weeks for each patient

SECONDARY OUTCOMES:
Rate of patients with DSC > 0.85 for other organs at risk (oral cavity, medullar canal, mandible,brain stem, larynx) | 7 weeks for each patient
Rate of patients with DSC > 0.85 for target volumes (clinical target volume, gross target volume, planning target volume) | 7 weeks for each patient
Time saving defined by the difference between standard recontouring time (manuel recontouring) and experimental recontouring time (Precise ART™ or Precise RTX™) | 7 weeks for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire Du Cancer Toulouse - Oncopole (Iuct-O), Toulouse, France